CLINICAL TRIAL: NCT06484478
Title: A Real-world Monitoring Project Exploring Day-to-day Physical Activity, Sleep, and Quality of Life in Individuals with Fabry Disease.
Brief Title: A Real-world Wearables Study in Fabry Disease.
Status: Recruiting | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Brunel University (Other)
Responsible Party: Sponsor
Other Study IDs: 320134
Record Dates: First submitted 2024-06-12; First posted 2024-07-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with Fabry disease
  Interventions: Other: Wearable technology monitoring

INTERVENTIONS:
Other: Wearable technology monitoring — Observational study (no intervention delivered)

SUMMARY:
Despite improvements in Fabry disease care in recent years, many patients still have poor outcomes. In addition to the many physical symptoms that patients can experience, the disease also places individuals at an increased risk of mental health conditions, such as anxiety and depression. Low physical activity levels and increased sedentary time are detrimentally associated with anxiety, depression and quality of life in the general population. Currently, no such research has been conducted in individuals with Fabry disease.

Data will consist of: (1) information from hospital medical records, (2) patient reported outcomes collected via questionnaires, and (3) measurements from a clinical-grade wearable device.

Individuals with Fabry disease aged 18 years or above will be considered for eligibility screening.

DETAILED DESCRIPTION:
Trial assessments:

Baseline questionnaires

Baseline questionnaires will include the Hospital Anxiety and Depression Scale (HADS) and the EuroQol 5-dimension questionnaire (EQ-5D-5L). This will be administered via Qualtrics.

Thigh-worn device (activPAL)

Participants will attach the activPAL device to their anterior thigh for 8 days and continue their usual daily behaviour throughout the week. This will measure sitting, standing, stepping and sleep time. This device is accompanied by a hard copy daily diary, where participants will be asked to input the time they wake up, they get out of bed, they get into bed, and when they go to sleep.

Clinical data

Data from medical records will include disease phenotype and clinical severity including mutation type, lyso-Gb3, left ventricular mass index and diastolic dysfunction. Such data will be sourced from electronic patient records. Mainz Severity Score Index, and its age-adjusted score will be calculated from data on electronic patient records. These will be collected retrospectively from the previous 12 months upon enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fabry disease documented by genotyping and/or enzymatic analysis.
* Resident in the UK.
* Aged 18 years and over.
* Capable of providing informed consent.
* Physically able to stand and ambulate independently.

Exclusion Criteria:

* A known allergy to any materials in the wearable device.
* Not able to have or use a wearable.
* Taking part in an interventional study which would preclude real-world data collection.
* Unable to communicate in English to a sufficient level to permit engagement in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Fabry disease who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life - via EuroQol five-dimension questionnaire (EQ-5D-5L). | Baseline
  Quality of life measured using the self-report EuroQol five-dimension questionnaire (EQ-5D-5L). The questionnaire is comprised of five dimensions which are each divided into five levels of severity i.e. 1 = no problem, 2 = slight problems, 3 = moderate problems, 4 = severe problems, and 5 = unable to/extreme problems. A five-digit health state score is then found by combining the levels of severity for each dimension i.e. 11111 is the best health state and 55555 is the worst health state.

SECONDARY OUTCOMES:
Anxiety | Baseline
  Anxiety measured using the self-report Hospital Anxiety and Depression Scale (HADS) questionnaire. HADS has 14 questions which measure anxiety (7 questions) and depression (7 questions). Each question is scored from 0 to 3 and total scores for anxiety (out of 21) and depression (out of 21) are calculated. Scoring is as follows: 0 - 7 = normal, 8 - 10 = borderline abnormal and 11 - 21 = abnormal.
Depression | Baseline
  Depression measured using the self-report Hospital Anxiety and Depression Scale (HADS) questionnaire. HADS has 14 questions which measure anxiety (7 questions) and depression (7 questions). Each question is scored from 0 to 3 and total scores for anxiety (out of 21) and depression (out of 21) are calculated. Scoring is as follows: 0 - 7 = normal, 8 - 10 = borderline abnormal and 11 - 21 = abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No